CLINICAL TRIAL: NCT02488252
Title: Semi-individualised Chinese Medicine Treatment as an Adjuvant Management for Diabetic Nephropathy - A Pilot add-on, Randomised, Controlled, Multi-centre, Open-label Pragmatic Clinical Trial
Brief Title: Semi-individualised Chinese Medicine Treatment as an Adjuvant Management for Diabetic Nephropathy
Acronym: SCHEMATIC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: School of Chinese Medicine, The University of Hong Kong (Unknown)
Responsible Party: Principal Investigator, Sydney CW TANG, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DN-CM-1
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Nephropathies
Keywords: Chinese Medicine; ACEI; ARB; Pragmatic trial
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard medical care (Active Comparator): Angiotensin converting enzyme inhibitor or angiotensin receptor blocker and oral hypoglycemic agents or insulin at stable dose
  Interventions: Drug: Routine medical care (active comparator)
- Chinese Medicine on top of standard medical care (Experimental): Semi-individualised Chinese Medicine treatment on top of standard medical care The treatment plan consists of 5 different formulas and will be prescribed to patients categorised to 5 subgroups according to clinical manifestation. Patients having multiple manifestations that fit more than 1 subgroup will not be included.
  Minor adjustment of the medication will be allowed and determined by the Chinese Medicine practitioner to reflect actual clinical practice. Dosage will follow strictly the China Pharmacopeia.
  A: spleen and kidney Qi deficiency, B: spleen and kidney Yang deficiency, C: spleen and kidney Qi and Ying deficiency, D: liver and kidney Ying deficiency, E: Ying and Yang deficiency
  Rehmannia-6 decoction: Wolfiporia cocos, Rehmannia glutinosa, Common macrocarpium Fruit, Dioscorea opposita , Paeonia suffruticosa Andr., Oriental waterplantain rhizome
  Rehmannia-8 decoction: Radix Aconiti Lateralis preparata, Cinnamomum cassia Presl, Rehmannia-6 decoction
  Interventions: Drug: Semi-individualised Chinese Medicine treatment; Drug: Routine medical care (active comparator)

INTERVENTIONS:
Drug: Semi-individualised Chinese Medicine treatment — A: Panax ginseng, Atractylodes macrocephala, Pinellia ternate, Pericarpium citri reticulatae, Herba Pogostemonis, Glycyrrhiza uralensis, Rehmannia-6 decoction
  B: Cortex magnoliae officinalis, Atractylodes macrocephala, Common Floweringquince Fruit, Common Vladimiria Root, Tsaoko Amomum Fruit, Palmae Fruit, Radixaconiti laterlis perparata, Zingiber officinale Rosc., Glycyrrhiza uralensis, Rehmannia-8 decoction
  C: Root of Pilose Asiabell, Astragalus membranaceus, Rehmannia glutinosa, Common Macrocarpium Fruit, Dioscorea opposita , Barbary Wolfberry Fruit, Cortex eucommiae, Chinese Angelica, Glycyrrhiza uralensis
  D: Rehmannia-6 decoction, Fructus Ligustri Lucidi, Yerbadetajo Herb
  E: Rehmannia-8 decoction, Fructus Ligustri Lucidi, Yerbadetajo Herb
  Arms: Chinese Medicine on top of standard medical care
Drug: Routine medical care (active comparator) — Angiotensin converting enzyme inhibitor or angiotensin receptor blocker at stable dose

SUMMARY:
This study aims to explore the effect of an adjuvant semi-individualized Chinese medicine treatment plan on type 2 diabetic patients with stages 2 to 3 chronic kidney disease and macroalbuminuria. This study will collect preliminary data on treatment effect, variance, recruitment rate and attrition rate for the planning of a subsequent clinical trial.

DETAILED DESCRIPTION:
This will be an open-label randomised parallel pilot clinical trial.

Sample size justification The sample size is calculated based on the target control of inflation factor. In order to be 95% confident (two-sided) that the subsequent main study actually achieves a power of 80% with nominal power set at 90% (i.e., a 10% power forfeit), the inflation factor should be less than 1.15.

At IF = 1.15, a sample size of 80 is therefore needed to have 95% one-sided confidence that the main study will achieve at least the nominal power to test the hypothesis that an add-on of the whole Chinese medicine treatment plan could be more effective in stabilising the glomerular filtration rate among diabetic nephropathy patients when compared to having just routine care.

For subgroup analysis, a sample size of 25 patients per each subgroup could achieve 80% one-sided confidence that the effect of stabilising glomerular filtration rate is different within subgroups of similar CM clinical pattern.

With 5 subgroups, a sample size of 148 patients is needed in this pilot trial to allow a 15% attrition rate.

Data management A trial management committee (TMC) formed by Principal Investigator, Co-Investigator and Research Assistant will centralise all the data of the trial. Chinese Medicine Practitioner and Research Assistant will collect, clean and send the data of patients to TMC on a daily basis. Questionnaires on clinical presentation and Chinese Medicine diagnosis will be sent, collected and cleaned by TMC directly daily by Research Assistant. If there is no response from the patients after 30 days of the last contact, Research Assistant will follow up and call the patients. All data will be double entered to computer and cleaned before analysis to prevent data entry errors. All transfer of data will include encryption and follow the guidelines by European Directive on Good Clinical Practice and adhere to Data Protection Act to protect the patients' confidentiality. TMC will have regular meetings monthly with experts to discuss the progress of the trial.

Data analysis Missing values, if any, will be imputed with regression. Patient without a postrandomisation assessment for a particular efficacy endpoint will be excluded from the analysis of that endpoint.

Regression analyses will be used to compare the adjusted mean of estimated GFR, UACR, HbA1c, FBG, FGF-23, MCP-1 and Cystatin C at week 48 between 1) the combination of all intervention groups and combination of all control groups, 2) individual treatment subgroup and its matching control group , and 3) different control groups with the corresponding baseline values as covariates. Change score analysis will be supplemented.

To minimise Type I error inflation, the analysis will follow a hierarchical approach in the order of 1) individual treatment subgroup versus its control subgroup, 2) combination of all intervention groups versus the combination of all control groups as to avoid Type I error inflation. The primary outcomes are the change of GFR and UACR.

Subgroup analysis will be performed for CKD stage 2 and 3 separately. Sensitivity analyses will be performed for 1) missing data imputed with regression, 2) missing data imputed with last-observation-carried-forward (LOCF) and 3) per protocol drop out of patient.

The adverse events will be analysed in a narrative manner. The percentage of all adverse events and the rate of attrition due to adverse events will be compared between intervention groups and control groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes for at least 5 years;
* with an estimated glomerular filtration rate (GFR) ≥30 ˂90 mL/min/1.73m2 confirmed with repeat testing over three or more months calculated by the abbreviated MDRD study equation;
* persistent macroalbuminuria with spot urine albumin-to-creatinine ratio (UACR) ≥ 300 mg/g confirmed by at least 2 out of 3 consecutive first morning void urine samples;
* on stable dose of anti-diabetic drug including insulin for 12 weeks;
* on stable dose of angiotensin-converting-enzyme inhibitor or angiotensin receptor blocker for 12 weeks; and
* willing and able to give written informed consent

Exclusion Criteria:

* with known history of glomerulonephritis, polycystic kidney disease, systemic lupus erythematosus, any suggestive evidence of nondiabetic glomerulopathy;
* with known history of kidney transplant;
* with concurrent severe disorders of heart, brain, liver, and hematopoietic system, tumor and mental disorder;
* with deranged liver function;
* poorly controlled blood pressure;
* with known history of intolerance or malabsorption of oral medications;
* with uncontrollable urinary infection;
* experiencing pregnancy; or
* participating in other clinical trial within 30 days

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in estimated GFR | From baseline to 48 weeks after treatment
  Efficacy and safety
Change in spot urine albumin-to-creatinine ratio | From baseline to 48 weeks after treatment
  Efficacy and safety

SECONDARY OUTCOMES:
Change in fasting blood glucose (FBG) | From baseline to 48 weeks after treatment
Change in glycated haemoglobin (HbA1c) | From baseline to 48 weeks after treatment
Change in urinary Cystatin C | From baseline to 48 weeks after treatment
Change in urinary nephrin | From baseline to 48 weeks after treatment
Change in serum fibroblast growth factor 23 (FGF-23) | From baseline to 48 weeks after treatment
Change in urinary monocyte chemotactic protein 1 (MCP-1) | From baseline to 48 weeks after treatment
Change in urinary transforming growth factor beta-1 (TGF-β1) | From baseline to 48 weeks after treatment
Change in urinary vascular endothelial growth factor (VEGF) | From baseline to 48 weeks after treatment
Change in serum brain natriuretic peptide (BNP) | From baseline to 48 weeks after treatment
Change in fasting serum insulin | From baseline to 48 weeks after treatment
Change in serum C-peptide | From baseline to 48 weeks after treatment
Rate of CKD stage transition | From baseline to 48 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sydney CW TANG, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chan KW, Kwong ASK, Tan KCB, Lui SL, Chan GCW, Ip TP, Yiu WH, Cowling BJ, Taam Wong V, Lao L, Feng Y, Lai KN, Tang SCW. Add-on Rehmannia-6-Based Chinese Medicine in Type 2 Diabetes and CKD: A Multicenter Randomized Controlled Trial. Clin J Am Soc Nephrol. 2023 Sep 1;18(9):1163-1174. doi: 10.2215/CJN.0000000000000199. Epub 2023 Jun 12. PMID 37307005
- [Derived] Chan KW, Ip TP, Kwong AS, Lui SL, Chan GC, Cowling BJ, Yiu WH, Wong DW, Liu Y, Feng Y, Tan KC, Chan LY, Leung JC, Lai KN, Tang SC. Semi-individualised Chinese medicine treatment as an adjuvant management for diabetic nephropathy: a pilot add-on, randomised, controlled, multicentre, open-label pragmatic clinical trial. BMJ Open. 2016 Aug 5;6(8):e010741. doi: 10.1136/bmjopen-2015-010741. PMID 27496229